CLINICAL TRIAL: NCT02603770
Title: A Single Site, Randomized Open Label Cross-Over Study to Compare Pharmacokinetic Profiles (PK) of XueZhiKang (XZK) Capsules Versus Lovastatin Tablets in Healthy Male Volunteers
Brief Title: Compare Pharmacokinetic(PK) Profiles of XZK vs Lovastatin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LY02405/CT-USA-102
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Lipid Metabolism Disorder
MeSH Terms: conditions — Lipid Metabolism Disorders | interventions — xuezhikang; Lovastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XueZhiKang (XZK) (Experimental): XueZhiKang (XZK) 1200 mg
  Interventions: Drug: XueZhiKang
- Lovastatin (Active Comparator): Lovastatin 20 mg
  Interventions: Drug: Lovastatin

INTERVENTIONS:
Drug: XueZhiKang
  Other Names: XZK
  Arms: XueZhiKang (XZK)
Drug: Lovastatin
  Other Names: Mevacor
  Arms: Lovastatin

SUMMARY:
The objective of this study is to compare laboratory tests profiles of a botanic drug XueZhiKang (XZK) 300 mg capsules versus a marketed drug Lovastatin 20 mg tablets in healthy male volunteers between 18 and 50 years of age.

DETAILED DESCRIPTION:
Twenty (20) healthy male subjects will be enrolled and assigned to either XZK group or Lovastatin group at a 1:1 ratio at one site in the USA.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent and complying with study procedures;
* Male subjects between the ages of 18 and 50 years, inclusive;
* Considered healthy by the PI, based on a detailed medical history, physical examination, clinical laboratory tests, 12-lead ECG and vital signs;
* Nonsmoker, defined as not having smoked or used any form of tobacco in more than 6 months before screening;
* Body Mass Index (BMI) of 19 to 32 kg/m2 inclusive and body weight not less than 50 mg;
* Willing and able to adhere to study restrictions and to be confined at the clinical research center.

Exclusion Criteria:

* Clinically significant past history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity;
* History or presence of malignancy other than adequately treated basal cell skin cancer;
* Clinically relevant illness within one month prior to the screening visit or at screening visit that may interfere with the conduct of this study;
* Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) or hepatitis C antibody;
* A history of seizure. However, a history of febrile seizure is allowed;
* A hospital admission or major surgery within 30 days prior to screening;
* Participation in any other investigational drug trial within 30 days from the last dosing of other trials to screening;
* A history of prescription drug abuse, or illicit drug use within 6 months prior to screening;
* A history of alcohol abuse according to medical history within 6 months prior to screening;
* A positive screen for alcohol, drugs of abuse;
* Tobacco use within 6 months prior to screening based on subject report;
* Subjects with hypersensitivity to lipid-lowering agents;
* Subjects who have participated in a previous clinical study of XZK;
* An unwillingness or inability to comply with food and beverage restrictions during study participation;
* Donation or blood collection of more than 1 unit (approximately 450 ml) of blood (or blood products) or acute loss of blood during the 90 days prior to screening;
* Use of prescription or over-the-counter (OTC) medications, and herbal (including St. John's Wort, herbal teas, garlic extracts) within 14 days prior to dosing (Note: Use of acetaminophen at < 3g/day is permitted until 24 hours prior to dosing).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
AUC for the Pharmacokinetics (PK) of XZK | 12 days
  PK Samples drawn at 0 (within 30 minutes prior to dosing), 0.5, 1,2,3,4 (+/- 5 min), 6,8,12 and 24 hour (+/- 15 min) after dosing on Day 1 and Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Simon LI, M.D., Study Chair — Luye Pharma
Locations (1):
- NRC Research Institute, Orange, California, United States